CLINICAL TRIAL: NCT05298670
Title: Drug Repurposing Using Metformin for Improving the Therapeutic Outcome in Multiple Sclerosis Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: German University in Cairo (Other)
Responsible Party: Principal Investigator, Mohamed Youssef Elsayed, Research assistant in Clinical Pharmacology and Pharmacogenomics Research Gruop, German University in Cairo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSMet
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Metformin; Tablets; Interferon beta-1a

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Cidophage®) and Interferon Beta 1 a (Rebiff ® 44mcg or Avonex ®) (Experimental): Metformin 1000 mg (Cidophage® 1000 mg tablets, CID, Giza, Egypt) tablet twice daily for 6 months as add on therapy with Interferon beta 1 a (Rebiff ® 44mcg or Avonex ®).
  Interventions: Drug: MetFORMIN 1000 Mg Oral Tablet; Drug: Interferon beta-1a
- Interferon beta 1 a (Rebiff ® 44mcg or Avonex ®) (Active Comparator): Interferon beta 1 a (Rebiff ® 44mcg or Avonex ®)
  Interventions: Drug: Interferon beta-1a

INTERVENTIONS:
Drug: MetFORMIN 1000 Mg Oral Tablet — Antidiabetic agent used to treat type 2 diabetes, and to prevent type 2 diabetes.
  Other Names: Cidophage ®1000 mg tablets, CID, Giza, Egypt) tablet and Rebiff ® 44mcg or Avonex®
  Arms: Metformin (Cidophage®) and Interferon Beta 1 a (Rebiff ® 44mcg or Avonex ®)
Drug: Interferon beta-1a — Disease Modifying Therapies (DMTs)
  Other Names: Rebiff ® 44mcg or Avonex®

SUMMARY:
This study aims to evaluate the effect of Metformin as add- on therapy for improving the outcome in RRMS patients.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune-mediated neurodegenerative disease of the central nervous system characterized by inflammatory demyelination with axonal transection. Worldwide, there are about 2.3 million MS patients. Women are twice as likely to have MS as men. MS typically presents in young adults (mean age of onset, 20-30 years) and can lead to physical disability, cognitive impairment, and decreased quality of life.

The four main types of multiple sclerosis are clinically isolated syndrome (CIS), relapsing-remitting MS (RRMS), secondary progressive MS (SPMS), and primary progressive MS (PPMS). This research focuses on RRMS as it is the most common type (80%- 85%).

Elevated level of Interleukins, and oxidative stress parameters are associated with MS pathology which exaggerated the myelin destruction, axonal degradation, and inflammatory cascade.

Metformin has a global safety record, is well-tolerated by the majority of patients and is used by roughly 125 million people worldwide, so a lot of studies inside and outside Egypt investigates their potential effect in different disorders as neurodegenerative diseases and cancer. Despite the prevalence of animal studies which explored Metformin neuroprotective effects by decreasing T- helper cells (Th 1 and Th 17) and improving Oligodendrocyte progenitor cell responsiveness to induce remyelination, clinical trials are still insufficient which motivate us to investigate the promising effect of Metformin as add-on treatment in RRMS patients

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years at time of signing informed consent form.
* Relapsing- remitting multiple sclerosis as per the McDonald 2017 criteria, including an MRI brain satisfying the 2017 radiological criteria.
* Full-field visual evoked potential (VEP) P100 latency in at least one eye of ≥118 ms.
* Kurtzke EDSS step 0.0 - 6.0.
* At the time of screening, being treated with a stable dose for at least 6 months of a category 1 multiple sclerosis DMT or for at least 2 years with a category 2 DMT.

Exclusion Criteria:

* People taking medication for Diabetes Mellitus at screening.
* Female participants who are pregnant, lactating, planning pregnancy, or unwilling to use reliable contraception during the trial.
* Significant liver impairment; alanine aminotransferase > 3 times the upper limit of normal.
* People suffering from congestive heart failure, chronic lung disease with hypoxia, and severe anemia.
* Patients with compromised renal function ((eGFR <60 mL/min/1.73m2) or coexistent hypoxic conditions should not be given metformin.
* Chronic or acute intake of large amounts of alcohol may potentiate the effect of metformin on lactate metabolism.
* Patients had been prescribed oral, intravenous, and intramuscular corticosteroids for one month prior to study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-28 (Estimated)

PRIMARY OUTCOMES:
Change in IL17 in both arms as measured by ELISA. | After 6 months
  Anti-inflammatory marker

SECONDARY OUTCOMES:
Percentage of Quality of Life deterioration in both arms measured by MSQOL-54. | After 6 months
  Assessment of quality of life for patients, The highest and lowest values refer to the satisfaction degree of patients
Change in IL22 in both arms as measured by ELISA. | After 6 months
  Anti-inflammatory marker
Malondialdehyde in both arms as measured by Colorimetric tests. | After 6 months
  Anti-oxidant marker
Degree of remyelination visualized by MRI, it depends on clinician's overview. | After 6 months
  Determination of T2 lesions
Degree of disability assessed by Expanded Disability Status Scale. | After 6 months
  Determination disability level (0 - 6), The lowest value means that it is best outcome and the highest value is the worst outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Nasser Institute for Research and Treatment, Cairo, Egypt

REFERENCES:
- [Background] Loma I, Heyman R. Multiple sclerosis: pathogenesis and treatment. Curr Neuropharmacol. 2011 Sep;9(3):409-16. doi: 10.2174/157015911796557911. PMID 22379455
- [Background] Browne P, Chandraratna D, Angood C, Tremlett H, Baker C, Taylor BV, Thompson AJ. Atlas of Multiple Sclerosis 2013: A growing global problem with widespread inequity. Neurology. 2014 Sep 9;83(11):1022-4. doi: 10.1212/WNL.0000000000000768. No abstract available. PMID 25200713
- [Background] Sormani MP, De Rossi N, Schiavetti I, Carmisciano L, Cordioli C, Moiola L, Radaelli M, Immovilli P, Capobianco M, Trojano M, Zaratin P, Tedeschi G, Comi G, Battaglia MA, Patti F, Salvetti M; Musc-19 Study Group. Disease-Modifying Therapies and Coronavirus Disease 2019 Severity in Multiple Sclerosis. Ann Neurol. 2021 Apr;89(4):780-789. doi: 10.1002/ana.26028. Epub 2021 Feb 9. PMID 33480077
- [Background] Pegoretti V, Swanson KA, Bethea JR, Probert L, Eisel ULM, Fischer R. Inflammation and Oxidative Stress in Multiple Sclerosis: Consequences for Therapy Development. Oxid Med Cell Longev. 2020 May 12;2020:7191080. doi: 10.1155/2020/7191080. eCollection 2020. PMID 32454942
- [Background] Negrotto L, Farez MF, Correale J. Immunologic Effects of Metformin and Pioglitazone Treatment on Metabolic Syndrome and Multiple Sclerosis. JAMA Neurol. 2016 May 1;73(5):520-8. doi: 10.1001/jamaneurol.2015.4807. PMID 26953870
- [Background] Triggle CR, Ding H. Metformin is not just an antihyperglycaemic drug but also has protective effects on the vascular endothelium. Acta Physiol (Oxf). 2017 Jan;219(1):138-151. doi: 10.1111/apha.12644. Epub 2016 Jan 13. PMID 26680745
- [Background] Sportelli C, Urso D, Jenner P, Chaudhuri KR. Metformin as a Potential Neuroprotective Agent in Prodromal Parkinson's Disease-Viewpoint. Front Neurol. 2020 Jun 12;11:556. doi: 10.3389/fneur.2020.00556. eCollection 2020. PMID 32595595
- [Background] Demare S, Kothari A, Calcutt NA, Fernyhough P. Metformin as a potential therapeutic for neurological disease: mobilizing AMPK to repair the nervous system. Expert Rev Neurother. 2021 Jan;21(1):45-63. doi: 10.1080/14737175.2021.1847645. Epub 2020 Dec 4. PMID 33161784
- [Background] Shi Q, Liu S, Fonseca VA, Thethi TK, Shi L. Effect of metformin on neurodegenerative disease among elderly adult US veterans with type 2 diabetes mellitus. BMJ Open. 2019 Jul 30;9(7):e024954. doi: 10.1136/bmjopen-2018-024954. PMID 31366635
- [Background] Dowling RJ, Goodwin PJ, Stambolic V. Understanding the benefit of metformin use in cancer treatment. BMC Med. 2011 Apr 6;9:33. doi: 10.1186/1741-7015-9-33. PMID 21470407
- [Background] Brown JR, Chan DK, Shank JJ, Griffith KA, Fan H, Szulawski R, Yang K, Reynolds RK, Johnston C, McLean K, Uppal S, Liu JR, Cabrera L, Taylor SE, Orr BC, Modugno F, Mehta P, Bregenzer M, Mehta G, Shen H, Coffman LG, Buckanovich RJ. Phase II clinical trial of metformin as a cancer stem cell-targeting agent in ovarian cancer. JCI Insight. 2020 Jun 4;5(11):e133247. doi: 10.1172/jci.insight.133247. PMID 32369446
- [Background] Ayoub R, Ruddy RM, Cox E, Oyefiade A, Derkach D, Laughlin S, Ades-Aron B, Shirzadi Z, Fieremans E, MacIntosh BJ, de Medeiros CB, Skocic J, Bouffet E, Miller FD, Morshead CM, Mabbott DJ. Assessment of cognitive and neural recovery in survivors of pediatric brain tumors in a pilot clinical trial using metformin. Nat Med. 2020 Aug;26(8):1285-1294. doi: 10.1038/s41591-020-0985-2. Epub 2020 Jul 27. PMID 32719487
- [Background] El-Khayat SM, Abouegylah M, Abdallah D, Geweil AG, Elenbaby AM, Zahra OS. The effect of metformin when combined with neoadjuvant chemotherapy in breast cancer patients. Med Oncol. 2021 Nov 5;39(1):1. doi: 10.1007/s12032-021-01599-3. PMID 34739637
- [Background] El-Fatatry BM, Ibrahim OM, Hussien FZ, Mostafa TM. Role of metformin in oxaliplatin-induced peripheral neuropathy in patients with stage III colorectal cancer: randomized, controlled study. Int J Colorectal Dis. 2018 Dec;33(12):1675-1683. doi: 10.1007/s00384-018-3104-9. Epub 2018 Jun 21. PMID 29931409
- [Background] Neumann B, Baror R, Zhao C, Segel M, Dietmann S, Rawji KS, Foerster S, McClain CR, Chalut K, van Wijngaarden P, Franklin RJM. Metformin Restores CNS Remyelination Capacity by Rejuvenating Aged Stem Cells. Cell Stem Cell. 2019 Oct 3;25(4):473-485.e8. doi: 10.1016/j.stem.2019.08.015. PMID 31585093
- [Background] Houshmand F, Barati M, Golab F, Ramezani-Sefidar S, Tanbakooie S, Tabatabaei M, Amiri M, Sanadgol N. Metformin-induced AMPK activation stimulates remyelination through induction of neurotrophic factors, downregulation of NogoA and recruitment of Olig2+ precursor cells in the cuprizone murine model of multiple sclerosis. Daru. 2019 Dec;27(2):583-592. doi: 10.1007/s40199-019-00286-z. Epub 2019 Oct 16. PMID 31620963
- [Background] Vickrey BG, Hays RD, Harooni R, Myers LW, Ellison GW. A health-related quality of life measure for multiple sclerosis. Qual Life Res. 1995 Jun;4(3):187-206. doi: 10.1007/BF02260859. PMID 7613530
- [Background] Abdallah MS, Alarfaj SJ, Saif DS, El-Naggar ME, Elsokary MA, Elsawah HK, Abdelsattar Zaki S, Wahsh EA, Abo Mansour HE, Mosalam EM. The AMPK modulator metformin as adjunct to methotrexate in patients with rheumatoid arthritis: A proof-of-concept, randomized, double-blind, placebo-controlled trial. Int Immunopharmacol. 2021 Jun;95:107575. doi: 10.1016/j.intimp.2021.107575. Epub 2021 Mar 24. PMID 33773207
- [Derived] Abdelgaied MY, Rashad MH, El-Tayebi HM, Solayman MH. The impact of metformin use on the outcomes of relapse-remitting multiple sclerosis patients receiving interferon beta 1a: an exploratory prospective phase II open-label randomized controlled trial. J Neurol. 2024 Mar;271(3):1124-1132. doi: 10.1007/s00415-023-12113-2. Epub 2023 Dec 9. PMID 38070031